CLINICAL TRIAL: NCT00005161
Title: Longitudinal Twin Study - Cohort Study of Blood Pressure
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1033; R01HL031010 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

SUMMARY:
To analyze the genetic and environmental contributions of juvenile hemodynamic determinants of blood pressure, including cardiac output and systemic vascular pressure, to adult cardiovascular risk.

DETAILED DESCRIPTION:
BACKGROUND:

Identifying individuals at a young age who are at risk for future development of hypertension in adult life is a public health issue of great importance. The imperfect nature of blood pressure tracking throughout childhood and adolescence, and the fact that the genes which determine blood pressure in childhood may not be the same ones which operate in adulthood make it clear that improved predicting models are needed. The twin-parent study design allowed testing more subtle genetic and environmental hypotheses than was possible with nuclear families or twins alone. The longitudinal component permitted an analysis of developmental changes in the genetic expression of the hemodynamic determinants of blood pressure. The inclusion of unlike sex twins permitted an analysis of the consistency of genetic and environmental effects across the sexes.

DESIGN NARRATIVE:

The longitudinal comparison of the cardiovascular responses of adolescent twins and their parents was initialed in 1983. Three cohorts of twin families were enrolled, each cohort beginning 18 months apart. Both monozygotic and dizygotic twins were included. Variables measured included demographics, family history, personality, blood pressure, anthropometry, stage of puberty, dynamic exercise, isometric exercise, psychological stress, echocardiography, genotyping, and lipid profiles. Each cohort revisited every 18 months.

A fourth cohort of 330 preadolescent twin pairs stratified by sex and zygosity was recruited from an established population-based twin registry. The hemodynamic determinants of blood pressure were assessed by non-invasive measurements of cardiac function including echocardiography and response to isometric and dynamic exercise. Zygosity was determined by questionnaire and confirmed by dermatoglyphic analysis and blood group tests. Anthropometric and hemodynamic measurements in the parents were compared to those in the children. The study included up to five sets of longitudinal measurements, thereby permitting an evaluation of whether the same or different genes operated at different ages encompassing pre-puberty, puberty, and post-puberty.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1983-08; Study Completion 1993-07

REFERENCES:
- [Background] van den Bree MB, Schieken RM, Moskowitz WB, Eaves LJ. Genetic regulation of hemodynamic variables during dynamic exercise. The MCV twin study. Circulation. 1996 Oct 15;94(8):1864-9. doi: 10.1161/01.cir.94.8.1864. PMID 8873661
- [Background] Nance WE. The relevance of twin studies to cardiovascular research. Prog Clin Biol Res. 1984;147:325-48. No abstract available. PMID 6377316
- [Background] Schieken RM: Exercise Study of Blood Pressure: A Predictor of Future Hypertension? In: NHLBI Workshop on Juvenile Hypertension, Loggie JHM, Horan M, Gruskin AB, et al (Eds.), Biomedical Information Corporation, NY, NY, 1984
- [Background] Schieken RM: Children's Blood Pressure. Report of 8th Ross Conference on Pediatric Research, Columbus Ohio: Ross Laboratories, 1985
- [Background] Corey LA, Eaves LJ, Mellen BG, Nance WE. Testing for developmental changes in gene expression on resemblance for quantitative traits in kinships of twins: application to height, weight, and blood pressure. Genet Epidemiol. 1986;3(2):73-83. doi: 10.1002/gepi.1370030203. PMID 3710139
- [Background] Eaves LJ, Long J, Heath AC. A theory of developmental change in quantitative phenotypes applied to cognitive development. Behav Genet. 1986 Jan;16(1):143-62. doi: 10.1007/BF01065484. No abstract available. PMID 3707482
- [Background] Schieken RM, Lauer RM, Clarke WR. Hemodynamics in childhood hypertension. Clin Exp Hypertens A. 1986;8(4-5):703-20. doi: 10.3109/10641968609046588. PMID 3757286
- [Background] Bodurtha JN, Schieken R, Segrest J, Nance WE. High-density lipoprotein-cholesterol subfractions in adolescent twins. Pediatrics. 1987 Feb;79(2):181-9. PMID 3808790
- [Background] Schieken RM. Measurement of left ventricular wall mass in pediatric populations. Hypertension. 1987 Feb;9(2 Pt 2):II47-52. doi: 10.1161/01.hyp.9.2_pt_2.ii47. PMID 3804400
- [Background] Martin NG, Clark P, Ofulue AF, Eaves LJ, Corey LA, Nance WE. Does the PI polymorphism alone control alpha-1-antitrypsin expression? Am J Hum Genet. 1987 Mar;40(3):267-77. PMID 3495177
- [Background] Hewitt JK, Eaves LJ, Neale MC, Meyer JM. Resolving causes of developmental continuity or "tracking." I. Longitudinal twin studies during growth. Behav Genet. 1988 Mar;18(2):133-51. doi: 10.1007/BF01067836. No abstract available. PMID 3377729
- [Background] Schieken RM, Moskowitz WB, Bodurtha J, Mosteller M, Eaves L, Nance W. Aortic stiffness: a new Doppler echocardiographic measure predictive of systolic blood pressure in children. J Am Coll Cardiol. 1988 Jun;11(6):1297-300. doi: 10.1016/0735-1097(88)90295-1. PMID 3367005
- [Background] Eaves LJ, Hewitt JK, Heath AC: The Quantitative Study of Human Developmental Change: A Model and its Limitations. 2nd International Conference on Quantitative Genetics, Sinauer Associates, 1988
- [Background] Schieken RM. Identification of high risk relatives for coronary heart disease. J Am Coll Cardiol. 1988 Oct;12(4):1110-3. doi: 10.1016/0735-1097(88)90487-1. PMID 2971084
- [Background] Schieken RM. Preventive cardiology: an overview. J Am Coll Cardiol. 1988 Oct;12(4):1090-1. doi: 10.1016/0735-1097(88)90481-0. No abstract available. PMID 3417981
- [Background] Schieken RM. The management of the family at high risk for coronary heart disease. Cardiol Clin. 1989 May;7(2):467-77. PMID 2659186
- [Background] Schieken RM, Eaves LJ, Hewitt JK, Mosteller M, Bodurtha JN, Moskowitz WB, Nance WE. Univariate genetic analysis of blood pressure in children (the Medical College of Virginia Twin Study). Am J Cardiol. 1989 Dec 1;64(19):1333-7. doi: 10.1016/0002-9149(89)90577-8. PMID 2686389
- [Background] Moskowitz WB, Mosteller M, Schieken RM, Bossano R, Hewitt JK, Bodurtha JN, Segrest JP. Lipoprotein and oxygen transport alterations in passive smoking preadolescent children. The MCV Twin Study. Circulation. 1990 Feb;81(2):586-92. doi: 10.1161/01.cir.81.2.586. PMID 2297864
- [Background] Bodurtha JN, Mosteller M, Hewitt JK, Nance WE, Eaves LJ, Moskowitz WB, Katz S, Schieken RM. Genetic analysis of anthropometric measures in 11-year-old twins: the Medical College of Virginia Twin Study. Pediatr Res. 1990 Jul;28(1):1-4. doi: 10.1203/00006450-199007000-00001. PMID 2377391
- [Background] Schieken RM. Left ventricular mass. Development versus disease. Circulation. 1990 Oct;82(4):1525-7. doi: 10.1161/01.cir.82.4.1525. No abstract available. PMID 2144801
- [Background] Fabsitz RR, Carmelli D, Hewitt JK. Evidence for independent genetic influences on obesity in middle age. Int J Obes Relat Metab Disord. 1992 Sep;16(9):657-66. PMID 1328090
- [Background] Schieken RM. Effects of childhood hypertension on the heart. The heart and hypertension. Child Nephrol Urol. 1992;12(2-3):128-32. No abstract available. PMID 1385756
- [Background] Goble MM, Mosteller M, Moskowitz WB, Schieken RM. Sex differences in the determinants of left ventricular mass in childhood. The Medical College of Virginia Twin Study. Circulation. 1992 May;85(5):1661-5. doi: 10.1161/01.cir.85.5.1661. PMID 1572024
- [Background] Goble MM, Schieken RM. Blood pressure response to exercise. A marker for future hypertension? Am J Hypertens. 1991 Nov;4(11):617S-620S. doi: 10.1093/ajh/4.11s.617s. PMID 1789943
- [Background] Implementation of hospital-based technology assessment. Int J Technol Assess Health Care. 1997 Summer;13(3):495. No abstract available. PMID 9308285
- [Background] Verhaaren HA, Schieken RM, Mosteller M, Hewitt JK, Eaves LJ, Nance WE. Bivariate genetic analysis of left ventricular mass and weight in pubertal twins (the Medical College of Virginia twin study). Am J Cardiol. 1991 Sep 1;68(6):661-8. doi: 10.1016/0002-9149(91)90361-n. PMID 1877484
- [Background] Bodurtha JN, Chen CW, Mosteller M, Nance WE, Schieken RM, Segrest J. Genetic and environmental contributions to cholesterol and its subfractions in 11-year-old twins. The Medical College of Virginia Twin Study. Arterioscler Thromb. 1991 Jul-Aug;11(4):844-50. doi: 10.1161/01.atv.11.4.844. PMID 2065038
- [Background] Moskowitz WB, Newkumet KM, Albrecht GT, Goble MM, Schieken RM. Case of steel versus steal: coil embolization of congenital coronary arteriovenous fistula. Am Heart J. 1991 Mar;121(3 Pt 1):909-11. doi: 10.1016/0002-8703(91)90208-y. No abstract available. PMID 2000759
- [Background] Newkumet KM, Goble MM, Young RB, Kaplowitz PB, Schieken RM. Altered blood pressure reactivity in adolescent diabetics. Pediatrics. 1994 Apr;93(4):616-21. PMID 8134217
- [Background] Schieken R. Premature atherosclerosis and familial hypercholesterolemia. Coron Artery Dis. 1993 Feb;4(2):126-32. doi: 10.1097/00019501-199302000-00002. No abstract available. PMID 8269204
- [Background] Austin MJ, Neale MC, Corey LA, Nance WE, Schieken RM, Brown JA. Common fragile site expression in lymphocytes from an individual mosaic for trisomy 8. Am J Med Genet. 1993 Mar 1;45(5):570-1. doi: 10.1002/ajmg.1320450509. PMID 8456825
- [Background] Schieken RM. Genetic factors that predispose the child to develop hypertension. Pediatr Clin North Am. 1993 Feb;40(1):1-11. doi: 10.1016/s0031-3955(16)38476-0. PMID 8417398
- [Background] Verhaaren HA, Schieken RM, Schwartz P, Mosteller M, Matthys D, Maes H, Beunen G, Vlietinck R, Derom R. Cardiovascular reactivity in isometric exercise and mental arithmetic in children. J Appl Physiol (1985). 1994 Jan;76(1):146-50. doi: 10.1152/jappl.1994.76.1.146. PMID 8175499
- [Background] Moskowitz WB, Mosteller M, Hewitt JK, Eaves LJ, Nance WE, Schieken RM. Univariate genetic analysis of oxygen transport regulation in children: the Medical College of Virginia Twin Study. Pediatr Res. 1993 Jun;33(6):645-8. doi: 10.1203/00006450-199306000-00022. PMID 8378126
- [Background] Moore WE, Burmeister JA, Brooks CN, Ranney RR, Hinkelmann KH, Schieken RM, Moore LV. Investigation of the influences of puberty, genetics, and environment on the composition of subgingival periodontal floras. Infect Immun. 1993 Jul;61(7):2891-8. doi: 10.1128/iai.61.7.2891-2898.1993. PMID 8514392
- [Background] Schieken RM. Why screen children for blood cholesterol levels? Ann Epidemiol. 1991 Nov;1(6):571-4. doi: 10.1016/1047-2797(91)90030-g. No abstract available. PMID 1669538
- [Background] Schieken RM. Effect of exercise on lipids. Ann N Y Acad Sci. 1991;623:269-74. doi: 10.1111/j.1749-6632.1991.tb43736.x. No abstract available. PMID 2042835